CLINICAL TRIAL: NCT04370860
Title: Determine the Optimal EGFR TKIs Treatment Strategies for Lung Adenocarcinoma Harboring EGFR Exon 19 Deletion Variants : the Clinical Analysis and Cell Lines Study
Brief Title: Optimal EGFR TKIs Treatment Strategies for Lung Adenocarcinoma Harboring EGFR Exon 19 Deletion Variants
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202002122RINC
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2021-06

CONDITIONS: EGFR Exon 19 Mutation; Tumor Progression
Keywords: epidermal growth factor receptor tyrosine inhibitor; lung adenocarcinoma
MeSH Terms: conditions — Disease Progression; Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Biopsy tissue, DNA, RNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine the optimal EGFR TKIs treatment strategies for lung adenocarcinoma harboring EGFR exon 19 deletion variants

DETAILED DESCRIPTION:
RNA extraction: The investigators will extract total RNA from cell lysates by using Tri-reagent (Molecular Research Center, Inc., Cincinnati, Ohio) and an RNA Mini Kit (Qiagen, Hilden, Germany) according to the manufacturer's instruction. RNA obtained from the Mini Kit column will be eluted. The quantity and quality of the purified RNA will be evaluated using a NanoDrop ND-1000 spectrophotometer will be stored at -80 °C for further mutational analyses.

Data acquisition: The investigators will record and follow participants' clinical information, including ethnicity, age, gender, smoking status, histological types, lung cancer stage (the TNM status), metastatic sites, ECOG score, CT/CXR imaging, chemotherapy or radiation treatment at the time of diagnosis of lung cancer and through the entire clinical courses. Specific marker such as TTF1, is used to ensure the diagnosis of primary lung tumor. Clinicopathologic stage assigns according to the seventh tumor-node-metastasis classification. The investigators assess the treatment responses according to the Response Evaluation Criteria in Solid Tumors (RECIST) using the unidimension method, and record the best response achieved per treatment. Treatment response, progression-free survival, and overall survival are recorded prospectively for further analysis.

Statistical analysis: All categorical variables will be analyzed with Pearson's χ² test, except where a small size required the use of Fisher's exact test. The progression-free survival curve and overall survival will be plotted by the Kaplan-Meier method and compared by the log-rank test. Multivariate analysis for overall survival will be performed using the Cox's proportional hazards model. Two-sided p-values of less than 0.05 is considered significant. All analyses will be performed using SPSS software (version 16.0 for Windows; SPSS Inc.).

ELIGIBILITY:
Inclusion Criteria:

* Patients have signed the informed consent (201103013RC and 201111039RIC) before 2019/12/31 and authorized the Institutional Review Board of Nation Taiwan University Hospital to review the new study for approving the usage of residual specimens.
* The residual samples from various sources, including surgical tissues, computed tomography (CT)-guided needle aspiration and/or biopsy, echo-guided needle aspiration and /or biopsy, bronchoscopic biopsy or brushing, bronchoalveolar lavage (BAL), endobronchial ultrasound guided needle aspiration, and lymph node aspiration, and pleural effusion specimens. The samples will be collected at the time of diagnostic procedure performed. All patients should sign an informed consent for purpose of using samples for molecular genetic testing.
* 1000 residual specimens will be used for the study.

Exclusion Criteria:

* Patients didn't sign the informed consent (201103013RC, 201111039RIC)
* The residual specimens are not qualified.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: only citizens of Taiwan will be enrolled.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Tumor size measurement for evaluating tumor progression | "up to 5 years," "from date of treatment (EGFR TKIs) until the date of first documented progression
  Tumor size is recorded using CT scan before the first day of of treatment and routine CT scan image is captured at each cycle of treatment to evaluate the growth of tumor.
  According to RECIST (The Response Evaluation Criteria in Solid Tumors), tumor progression will be assigned based on (1) a sum measurement of original target lesions that has increased more than 20%, (2) the reappearance of the original target lesions, (3) appearance of new lesions, and (4) a new lymph node metastatic lesion which is more than 10mm in diameter. Statistically, patients will be divided into several groups according to Exon 19 deletion variants, which is detected before the first day of treatment. The clinicopathologic characteristics (sex, age, smoking history) will be enrolled in multivariate analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan